CLINICAL TRIAL: NCT02039661
Title: Effect of Lidocaine Spray for Pain Relief During Endometrial Biopsy: a Randomized, Double-blind, Placebo-controlled Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kayseri Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Gökhan Açmaz, MD, Kayseri Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Gookhan
Record Dates: First submitted 2014-01-16; First posted 2014-01-17 (Estimated); Last update posted 2014-01-17 (Estimated); Status verified 2014-01

CONDITIONS: Pain
Keywords: Curettage;; Pain Score
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lidocaine Spray (Active Comparator)
  Interventions: Drug: Lidocaine Spray
- Placebo (Placebo Comparator): These patients received placebo spray.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lidocaine Spray — These patients received 2 puff lidocaine spray
  Arms: Lidocaine Spray
Drug: Placebo
  Arms: Placebo

SUMMARY:
The effect of lidocaine spray on pain relief during endometrial sampling.

DETAILED DESCRIPTION:
The study population will comprise women with abnormal uterine bleeding who will be scheduled for endometrial sampling or women who will have control biopsies before surgery due to other pathologies. We have two groups; the first group consisted of patients who receive lidocaine spray. The second group consisted of patients who receive placebo spray. Patients will be asked to rate their pain level on a standard continuous 100-mm VAS to quantify the pain. Pain scoring will be performed at 3 different time points: immediately before to the procedure, during the procedure(immediately following the removal of the speculum from the vagina at the end of the endometrial sampling, the patients will be asked to score their pain level experienced during the procedure), and 15 minutes after the procedure.

We will document the patients' demographics and medical information. All procedures will be performed by a single operator and the same team to avoid possible operator-dependent pain factors (counseling, patient preparation, attitude and operative steps during operation, moral and psychological support).

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years no allergy Patients with abnormal uterine bleeding

Exclusion Criteria:

* cervical stenosis myoma uteri pregnancy miscarriage chronic pelvic pain dysmenorrhea

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2013-11; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Pain Score | 3 months
  Patients were asked to rate their pain level on a standard continuous 100-mm VAS to quantify the pain. Pain scoring was performed at 3 different time points: immediately before to the procedure, during the procedure (immediately following the removal of the speculum from the vagina at the end of the endometrial sampling, the patients were asked to score their pain level experienced during the procedure), and 15 minutes after the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Gökhan Açmaz, MD, Principal Investigator — Kayseri Education and Research Hospital of Medicine
Locations (1):
- Kayseri Education and Research Hospital of Medicine, Kayseri, Turkey (Türkiye)